CLINICAL TRIAL: NCT01466452
Title: Antiplatelet Effect of Low Doses of Aspirin Taken Every 12 Hours in Patients Undergoing Coronary Artery Bypass Graft and/or Aortic Valve Surgery
Acronym: ASABYVALV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Catholic University, Italy (Other); University of Chieti (Other)
Responsible Party: Principal Investigator, Alessandro Parolari, Assistant Professor of Cardiac Surgery, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: S181/211
Record Dates: First submitted 2011-10-20; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aspirin 100 (Active Comparator)
  Interventions: Drug: Aspirin
- Aspirin 200 (Active Comparator)
  Interventions: Drug: Aspirin
- Aspirin 100 x 2 (Active Comparator)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — single-dose aspirin in 100 mg 1 tablet every 24 hours
  Arms: Aspirin 100
Drug: Aspirin — single-dose aspirin 200 mg 1 tablet every 24 hours
  Arms: Aspirin 200
Drug: Aspirin — double-dose aspirin 100 mg 1 tablet every 12 hours
  Arms: Aspirin 100 x 2

SUMMARY:
This study is a randomized open label study that implies the administration of asprin according to three different regimens.

The aims of the study are:

* to establish whether coronary artery bypass surgery and / or aortic valve replacement surgery with bioprostheses is associated with changes in the rate of platelet regeneration that can reduce the effectiveness of aspirin administered at a dose of 100mg/die in terms of inhibition of platelet biosynthesis of thromboxane A2.
* to determine whether these patients need a different (shorter) interval of administration in order to completely and permanently inhibit the platelet COX-1.

The endpoints of this study are:

- To evaluate the changes in the levels of TXB2 and 12-HETE in serum at 12 and 24 hours after administration of aspirin and the changes in the levels of 11-dehydro TXB2 urinary 8-iso-PGF2 alpha urinary, 2-3 dinor-6-chetoPGF1 alpha, Verify-NOW Aspirin, platelets crosslinked at 12 and 24 hours after administration of aspirin

ELIGIBILITY:
Inclusion Criteria:

* informed consent of the study signed
* coronary artery bypass graft and / or aortic valve replacement surgery with bioprostheses
* age between 55 and 80
* ejection fraction > 30%.

Exclusion Criteria:

* excessive bleeding (> 1000mL / 6 h) or the need of re operation for bleeding
* perioperative myocardial infarction
* stroke or renal failure requiring dialysis and need waiting for post-operative anticoagulation
* patients undergoing coronary artery bypass grafting procedure as a consequence of failed percutaneous coronary intervention
* patients undergoing off-pump coronary artery bypass graft
* overt kidney or liver disease
* therapies that influence the coagulation
* fertile women

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
change in the levels of TXB2 in serum at 12 and 24 hours after administration of aspirin | one year
change in the levels of 12-HETE in serum at 12 and 24 hours after administration of aspirin | one year

SECONDARY OUTCOMES:
change in the levels of 11-dehydro TXB2 urinary at 12 and 24 hours after administration of aspirin | one year
change in the levels of 8-iso-PGF2 alpha urinary at 12 and 24 hours after administration of aspirin | one year
change in the levels of 2-3 dinor-6-chetoPGF1 alpha at 12 and 24 hours after administration of aspirin | one year
change in the levels of Verify-NOW Aspirin, platelets crosslinked at 12 and 24 hours after administration of aspirin | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, IRCCS, Milan, Milano, Italy